CLINICAL TRIAL: NCT03704324
Title: Incidence and Risk Factors of PostopeRativE Delirium in ICU in China
Acronym: PREDICt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018ZSLC08
Record Dates: First submitted 2018-09-01; First posted 2018-10-12 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Delirium; Intensive Care Psychiatric Disorder
Keywords: Incidence and profile; Risk factors; Prediction model
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative delirium (POD) is a common postoperative complication that can occur in patients of any age. POD brings great burden to patients and their families, as the following cognitive decline may persist for months to years to impede patients returning to previous life quality and employment. The PREDICt study aims to characterize the incidence and profiles of POD in ICU, and to find out risk factors, especially any are modifiable, and any have value for developing prediction model. Our final aim is to comprehensively and deeply explore the etiology of POD to guide prevention of delirium among postoperative patients.

DETAILED DESCRIPTION:
Delirium is an acute and fluctuating alteration of mental state characterized by a disturbance in attention, level of consciousness and cognition. Postoperative delirium (POD) is a common postoperative complication that can occur in patients of any age, from children to elderly. POD was proved to be associated with several worse outcome, including increased mechanically ventilated duration, hospital length of stay (LOS) and cost. Moreover, the each day with delirium is independently associated with an increased hazard of death by 10%. Although studies on delirium substantially increased in the past decade, many research gaps still exist in this area due to the heterogeneity of their results. First, the incidence varies broad range because the targeted population are different. In China, up to now, no large sample studies to investigate the incidence and risk factors of POD in ICU. Moreover, although there have been numerous studies exploring the potential risk factors of POD, most of them are still with inconclusive evidence. The Benzodiazepine use and blood transfusion administration are the only two modifiable factors with strong evidence. Hence, still needs further studies to focus on etiology of POD to find out modifiable and non-modifiable factors to verify the presumed factors. Since there is lack of effective treatments for POD, prevention remains the best strategy to cope with delirium. Predictive models that include delirium risk factors can guide us to early prevention of high risk patients. There were two high-quality studies on prediction models for ICU delirium, named PRE-DELIRIC model and E-PRE-DELIRIC model. However, both of the models are conducted in general ICU, did not fully consider the factors of surgery.

The PREDICt study aims to find out risk factors, especially any are modifiable, and any have value for developing prediction model. Our primary aim is to determine the incidence and severity of Post-Operative Delirium (POD) in ICU after surgery, and identify the associated outcomes and burdens of POD in ICU by evaluating the impact on postoperative outcome, ICU and hospital length of stay, medical expenses. Our secondary aim is to investigate the modifiable and non-modifiable risk factors for the occurrence of POD during ICU stay and develop delirium prediction model for ICU patients. Our final aim is to comprehensively and deeply explore the etiology of POD to guide prevention of delirium among postoperative patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18
* Surgical patients
* Admitted to ICU after surgery

Exclusion Criteria:

* Preoperative delirium or dementia patients
* Unable to fully participate in delirium testing, including blind, deaf, illiterate or inability to understand Chinese
* Undergoing surgery procedures do not require admission to SICU
* Transfer to SICU from wards after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged above 18 who are admitted to surgical SICUs after operation will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | up to 20 days postoperatively
  Investigators screen delirium by CAM-ICU twice a day, each time during day and night.
  Investigators defined patients have delirium if they had at least one positive screening during ICU stay.

SECONDARY OUTCOMES:
Severity of postoperative delirium | up to 20 days postoperatively
  Assess by CAM-ICU-7 if CAM-ICU is positive. Categorized as no delirium: 0-2, mild to moderate delirium: 3-5, and severe delirium: 6-7.
duration of postoperative delirium | up to 20 days postoperatively
  Defined as time (in days) from the first positive CAM-ICU until the beginning of two consecutive days of negative CAM-ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Yuxia Zhang, Principal Investigator — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol has been published in Journal of advanced nursing
Supporting Information: Study Protocol, SAP
Time Frame: Estimated from 2019
Access Criteria: Study protocol has been published in Journal of advanced nursing

REFERENCES:
- [Derived] Cai S, Cui H, Pan W, Li J, Lin X, Zhang Y. Two-stage prediction model for postoperative delirium in patients in the intensive care unit after cardiac surgery. Eur J Cardiothorac Surg. 2022 Dec 2;63(1):ezac573. doi: 10.1093/ejcts/ezac573. PMID 36579859
- [Derived] Wang H, Zhao QY, Luo JC, Liu K, Yu SJ, Ma JF, Luo MH, Hao GW, Su Y, Zhang YJ, Tu GW, Luo Z. Early prediction of noninvasive ventilation failure after extubation: development and validation of a machine-learning model. BMC Pulm Med. 2022 Aug 8;22(1):304. doi: 10.1186/s12890-022-02096-7. PMID 35941641